CLINICAL TRIAL: NCT05411445
Title: Study of Role of Blood Microvescicles and Exosomes in Patients With Graft Occlusion After Aortocoronary Bypass Surgery
Acronym: MVBYPASS
Status: Recruiting | Type: Observational
Sponsor: Maria Cecilia Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MCH 2022-01
Record Dates: First submitted 2022-06-01; First posted 2022-06-09 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Bypass Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronary artery bypass graft (CABG) surgery is still the standard treatment of coronary revascularization for patients with severe coronary artery disease (CAD). Graft patency, together with completeness of revascularization, is a major determinant of long-term outcome following CABG. The surgical procedure elicits a persistent systemic inflammatory response associated with the activation of the hemostatic system leading to perturbation of endothelial and vascular function and activation of platelets and leukocytes. All of these events are the main players responsible for the early and late graft failure in a significant percentage of patients.

DETAILED DESCRIPTION:
Circulating microvesicles (MVs) have received increasing attention during the last years as novel players in cardiovascular disease. MVs are small membrane vesicles involved in cell-to-cell communication acting as biological messengers. MVs of different origin are present in the circulation of healthy subjects, and their number increases in several pathological conditions contributing to the development, progression, and clinical outcome of diseases. They have been proposed as biomarkers of thrombosis, vascular injury, and inflammation in atherothrombosis and myocardial infarction, where elevated levels have been correlated with disease severity. Among the circulating MVs, those expressing phosphatidylserine are defined as procoagulant MVs. A subgroup of procoagulant MVs also express tissue factor (TF), the key activator of the blood coagulation cascade. These procoagulant MVs have a role in the prediction of cardiovascular events and are able to identify patients at high recurrence risk. Thus far, many studies have generated compelling data on the sensitivity of circulating MVs as biomarkers of cardiovascular disease progression and events. The usefulness of MVs in patients undergoing CABG, however, has only been tested in 1 study that highlighted their importance in surgical hemostasis. No information is so far available on the association between the amount or pattern of circulating MVs and CABG outcome.Thus, we carried out this study to investigate potential functional role of MVs and exosomes in graft occlusion based on their protein profile as well as their procoagulant potentia.l

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 40 and 80
* Ejection fraction> 30%
* coronary artery bypass surgery
* informed consent
* Willingness to carry out the follow-up visits and the assessments required by the protocol

Exclusion Criteria:

* emergency intervention
* changes in liver or kidney function
* changes in coagulation factors
* associated interventions (valve replacement, carotid endarterectomy)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective CABG ( coronary artery bypass graft )
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Confirmation and validation of the potential role of blood MV and exosomes as predictors of bypass occlusions | from 15 to 21 months

CONTACTS AND LOCATIONS:
Locations (1):
- MCH, Cotignola, Ravenna, Italy

IPD SHARING:
Plan to Share IPD: No